CLINICAL TRIAL: NCT06349174
Title: Safety and Efficacy of Endobronchial Valve for Bronchoscopic Lung Volume Reduction Surgery: a Prospective Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-valve-1
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Emphysema; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endobronchial valve group (Experimental): The patients would undergo bronchoscopic lung volume reduction surgery using the self developed endobronchial valve.
  Interventions: Procedure: bronchoscopic lung volume reduction surgery using endobronchial valve

INTERVENTIONS:
Procedure: bronchoscopic lung volume reduction surgery using endobronchial valve — The patients would undergo bronchoscopic lung volume reduction surgery using the self developed endobronchial valve.

SUMMARY:
The goal of this pliot study al is to preliminarily evaluate the effectiveness and safety of transbronchial lung volume reduction surgery using the self-devloped endobronchial valves for chronic obstructive pulmonary disease patients with emphysema phenotype . The main questions it aims to answer are:

Does self-devloped endobronchial valves improve the lung function、exercise capacity and symptons of participants? What surgery-related adverse events do participants have after transbronchial lung volume reduction surgery using the self-devloped endobronchial valves?

Participants will:

undergo transbronchial lung volume reduction surgery using the self-devloped endobronchial valves.

receive follow-up before surgery (baseline) and 3 days, 4 weeks, 12weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with chronic obstructive pulmonary disease based on GOLD diagnostic criteria;
* 2. Age range from 40 to 85 years old (including 40 and 85 years old);
* 3. BMI ≤ 35kg/m2;
* 4. 15% ≤ FEV1% pred ≤ 45%;
* 5. TLC>100% pred, RV>140% pred, and DLCO/red% ≥ 20%;
* 6. 100m ≤ 6WMD ≤ 500m after rehabilitation training;
* 7. Quit smoking for more than 4 months;
* 8. The evaluation result of pulmonary bypass ventilation function is negative;
* 9. Participants in this clinical trial requires the signing of an informed consent form by the individual or legal representative.

Exclusion Criteria:

* 1. Being pregnant or breastfeeding;
* 2. PaCO2>50mmHg and/or PaO2<45mmHg;
* 3. Obvious bronchiectasis or other infectious lung diseases;
* 4. Hospitalization due to pulmonary infection or acute exacerbation of COPD within the past 12 months prior to baseline assessment twice or more times;
* 5. Coagulation dysfunction, platelet count<60e+09/L;
* 6. Myocardial infarction or congestive heart failure within the past 24 weeks;
* 7. Previous lobectomy, LVRS or lung transplantation;
* 8. Anticoagulant therapy that cannot be stopped before surgery;
* 9. Uncontrolled pulmonary arterial hypertension (systolic pulmonary arterial pressure>45mmHg) or lungs diagnosed within the past 12 weeks Arterial hypertension;
* 10. Left ventricular ejection fraction (LVEF) within the past 12 weeks is less than 45%;
* 11. Pulmonary nodules that require intervention;
* 12. Patients participating in other clinical trials;
* 13. Individuals with other contraindications to bronchial operations;
* 14. Other circumstances that the researcher deems unsuitable for participation in this clinical trial.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change in FEV1 relative to baseline | 12 weeks after surgery
  The patient will undergo lung function tests.

SECONDARY OUTCOMES:
Percentage of subjects with FEV1 improvement ≥ 12% after bronchodilators | 12 weeks after surgery
  The patient will undergo lung function tests.
Percentage change in RV relative to baseline | 12 weeks after surgery
  The patient will undergo lung function tests, and residual volume (RV) will be recorded.
Percentage change in TLC relative to baseline | 12 weeks after surgery
  The patient will undergo lung function tests, and total lung capacity (TLC) will be recorded.
Percentage change in DLCO relative to baseline | 12 weeks after surgery
  The patient will undergo lung function tests, and the diffusing capacity for carbon monoxide (DLCO) will be recorded.
Percentage change in SGRQ score relative to baseline | 12 weeks after surgery
  The patient will receive a St.Georges respiratory questionnaire (SGRQ) questionnaire survey.
Percentage change in mMRC grade relative to baseline | 12 weeks after surgery
  The patient will receive a modified Medical Research Council (mMRC) questionnaire.
Percentage change in 6MWD relative to baseline | 12 weeks after surgery
  The patient will undergo 6-minute walk test, and 6-minute walk distance (6MWD) will be recored.
the incidence of surgical-related adverse events | 12 weeks after surgery
  The surgical-related adverse events refers to pneumothorax, valve displacement or shedding, granuloma formation and other surgical-related adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No